CLINICAL TRIAL: NCT01101672
Title: A Randomized Controlled Trial Comparing the Outcomes of Patients Who Undergo Single Port Laparoscopic Colectomy and Conventional Laparoscopic Colectomy for Colonic Neoplasia
Brief Title: Trial for Single Port Versus Conventional Laparoscopic Colectomy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Jensen Poon, Department of Surgery, University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW09-341
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Last update posted 2010-04-12 (Estimated); Status verified 2010-04

CONDITIONS: Colonic Polyps; Colonic Cancers
Keywords: Single port laparoscopic colectomy
MeSH Terms: conditions — Colonic Polyps; Colonic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single-port laparoscopic colectomy (Experimental)
  Interventions: Procedure: Single port laparoscopic colectomy
- Conventinal laparoscopic colectomy (Active Comparator)
  Interventions: Procedure: Conventional laparoscopic colectomy

INTERVENTIONS:
Procedure: Single port laparoscopic colectomy — Patients will be operated by using the technique of single port laparoscopic colectomy by surgeon with experiences and training in this procedure. Laparoscopic instruments will be inserted to perform the procedure through a multi-channel single port which is placed via transumbilical incision. The same transumbilical incision will be extended to 3-4cm for extraction of specimen.
  Arms: Single-port laparoscopic colectomy
Procedure: Conventional laparoscopic colectomy — Patient will be operated by techniques of conventional laparoscopic colectomy. A 10mm subumbilical incision is made for camera port, another 2-4 small incisions (5-10mm in size) will be made for placement of ports and insertion of laparoscopic instrument. A 3-4cm abdominal incision will be made for extraction of specimen.
  Arms: Conventinal laparoscopic colectomy

SUMMARY:
This study aims to compare the outcomes of patients who undergo single-port laparoscopic colectomy and conventional laparoscopic colectomy for colonic neoplasia (large polyp not amenable to endoscopic removal/ cancer) through a randomized controlled trial. After informed consent, patients will be randomized to have either conventional or single-port laparoscopic colectomy by a team of surgeons with good experience in laparoscopic colorectal surgery. Patients' demographic, operative detail and post-operative outcomes including operating time, blood loss, complications, pain score, analgesic requirement, resumption of gastrointestinal function and length of hospital stay will be recorded prospectively. The patients will be blinded to the type of treatment that they have received during the first three days after operation (post-operative pain and analgesic requirement will be recorded in these period). Patients will have long term up to record for cancer recurrence and survival.

The results of two groups of patients will be compared scientifically to assess if single-incision laparoscopic colectomy results in any difference in outcomes when compared to conventional laparoscopic colectomy.

DETAILED DESCRIPTION:
Conventionally laparoscopic surgery requires multiple abdominal wall incision for placement of ports and laparoscopic instrument to perform the operation. With the advancement of technology, laparoscopic surgery can now be performed through one special port which can accommodate several laparoscopic instruments to perform the operation and hence, require only one small 2-3cm incision through the umbilicus. This is commonly named as Single-incision Laparoscopic Surgery (SILS) or single-port laparoscopic surgery.

Compared to conventional laparoscopic surgery, SILS has the advantage of further reduction of post-operative wound pain because of only one small abdominal incision is required. The cosmetic result from SILS is also better because the only incision is made through the umbilicus which can hide the wound effectively after operation. After complete healing of the umbilical wound, the patient's abdomen could be visually 'scarless'.

There has been no study to compare the results of the new single-port laparoscopic colectomy to the conventional laparoscopic colectomy in the literature yet. In order to decide if this new technique should be recommended to more patients for treatment of colonic neoplasia, a formal study is required. We designed a patient blinded randomized controlled trial to investigate if there is any difference between these two laparoscopic colectomies.

The primary outcome to be measured is post-operative pain on coughing and analgesia consumption. The patients will be blinded to the type of treatment that they have received during the first three days after operation. During these three days, the post-operative pain score and analgesic requirement will be recorded independently by the Pain team who is also blinded to the type of procedure.

The secondary to be measured include operating time, blood loss, morbidities and mortality, cancer recurrence and patient survival in long term. The secondary outcomes will also be recorded prospectively and compared.

Definition of conversion:

Conversion to conventional is defined as the need to place additional port to aid the procedure during the single port laparoscopic colectomy Conversion to open is defined as(1) the need to perform conventional laparotomy in order to accomplish the procedure or (2) premature abdominal incision for colorectal dissection or vascular control during single port or conventional laparoscopic colectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven neoplastic disease of colon (large polyps not amenable to endoscopic removal or cancer)
2. Age >18 years
3. Informed consent obtained
4. American Society of Anesthesiologist class 1-3

Exclusion Criteria:

1. Evidence of local invasion on pre-operative imaging
2. Cancer of diameter greater than 5cm
3. Contraindication for laparoscopic surgery
4. Anticipated peritoneal adhesion from previous major abdominal surgery
5. Presence of bowel obstruction
6. Lesion in transverse colon or rectum
7. Anticipated high dependency unit or intensive care unit admission after operation

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2009-11; Primary Completion 2011-07 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain on coughing | The first three days after operation
  The patients will be blinded to the type of treatment that they have received during the first three days after operation. During these three days, the post-operative pain score on coughing and analgesic requirement will be recorded independently by the Pain team of Department of Anesthesia who is also blinded to the type of procedure.

SECONDARY OUTCOMES:
Operative blood loss and transfusion | Immediate peri-operative period
Operative morbidities and 30 days mortality | 30 days after operation
Length of hospital stay | Time from operation to discharge
Recurrence and survival for cancer patient | The expected time frame of follow up is 2 year and 5 five after operation

CONTACTS AND LOCATIONS:
Overall Officials: Wai L Law, MS, MBBS, Study Chair — Department of Surgery, University of Hong Kong
Locations (1):
- Department of Surgery, Queen Mary Hospital, University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Background] Law WL, Fan JK, Poon JT. Single-incision laparoscopic colectomy: early experience. Dis Colon Rectum. 2010 Mar;53(3):284-8. doi: 10.1007/DCR.0b013e3181c959ba. PMID 20173474
- [Background] Law WL, Fan JK, Poon JT. Single incision laparoscopic left colectomy for carcinoma of distal transverse colon. Colorectal Dis. 2010 Jul;12(7):698-701. doi: 10.1111/j.1463-1318.2009.02114.x. Epub 2009 Nov 6. PMID 19895602